CLINICAL TRIAL: NCT05692063
Title: Anomalous Aortic Origin of Coronary Artery: From Pathophysiology to Risk Stratification Through a Patient Specific Computational Simulation Model
Brief Title: Anomalous Aortic Origin of Coronary Artery
Acronym: AAOCA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Mauro Lo Rito, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: AAOCA
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Anomalous Aortic Origin of the Coronary Artery (AAOCA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project has several objectives ranging from clinical data analysis to computational simulations as listed below:

A) Clinical objectives:

1. Retrospective review of all patients with AAOCA treated surgically and followed medically at the IRCCS Policlinico San Donato aiming to identify risk factors for ischemia or sudden cardiac deaths.
2. Prospective follow-up of all enrolled patients, treated and followed, in adjunct to all the new patients referred aiming to follow across the years any potential rare adverse event (ischemia, angina event, sudden cardiac death).

B) Experimental objectives:

1. Retrieve morphological measurements from CT or MRI (de-identified) of the aortic root and the coronary vessels following the previous work of our group.
2. Construct a parametric model of the aortic root defined by population-based morphologic parameters to describe both healthy/diseased population.
3. Run solid mechanics simulation mimicking the movement of the aortic root in order to test configurations at more risk.
4. Reconstruct 3D surfaces representing the coronary vasculature from imaging for automatically perform the parameter estimation and run computational fluid dynamics simulations.

ELIGIBILITY:
Inclusion Criteria:

* All patients (adults and pediatrics) who have been diagnosed with an anomalous aortic origin of any of the coronary arteries (AAOCA) without any other congenital heart disease and diagnosed/referred or followed at the IRCCS Policlinico San Donato.

Exclusion Criteria:

* Patients with other major congenital heart disease with associated coronary artery origin anomalies will be excluded.

Patients with anomalous origin of the coronary artery from the pulmonary artery (ALCAPA or ARCAPA) will be excluded.

Patients women who are pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (adults and pediatrics) with diagnosis of anomalous aortic origin of coronary arteries
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
ischemia, angina event, sudden cardiac death | 10 years
  2. Creation of a prospective registry in which will be enrolled all patients already treated and followed in adjunct to all the new patients referred aiming to follow across the years any potential rare adverse event

SECONDARY OUTCOMES:
risk factors for ischemia or sudden cardiac deaths | 10 years
  1. Retrospective review of all patients with AAOCA treated surgically and followed medically at the IRCCS Policlinico San Donato aiming to identify risk factors for ischemia or sudden cardiac deaths.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No